CLINICAL TRIAL: NCT03454776
Title: The Effect of the Unloader One® Knee Brace on Symptoms in Patients With Knee Osteoarthritis
Brief Title: Unloader One Study on Knee Osteoarthritis Hässleholm Sweden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Sören Toksvig-Larsen, Associate professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orthosestudy
Record Dates: First submitted 2018-01-29; First posted 2018-03-06 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Two groups with same problem of osteoarthritis in knee
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Unloader One brace (Active Comparator): Patients receiving an active brace, Unloader One with active straps facilitating unloading of affected knee compartment
  Interventions: Device: Unloader One brace
- Placebo brace (Placebo Comparator): Patients receiving a dummy, lookalike or placebo brace without active straps that facilitate unloading of the affected knee compartment
  Interventions: Device: Placebo brace

INTERVENTIONS:
Device: Unloader One brace — A knee brace used to unload affected compartments in osteoarthritic knees
  Arms: Unloader One brace
Device: Placebo brace — A knee brace that feels and looks like Unloader One but without active straps facilitating unloading of the knee
  Arms: Placebo brace

SUMMARY:
The purpose of this study is to assess the effect of the Unloader one brace on the clinical symptoms of patients with knee osteoarthritis (OA) by comparing a functioning brace with a dummy.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of the Unloader one brace on the clinical symptoms of patients with knee OA by comparing a functioning brace with a dummy. The dummy will be manufactured by Össur and has the same look as the real brace, but lacks the fundamental tightening effect of the straps of the real brace (an insert of elastic bands assures this), thereby nullifying its unloading capabilities. In a recent trial by Dr. Ingvarsson, the brace seemed to lessen the pain from knee OA, but no randomised, controlled studies have been conducted. This is mandatory if the effect of the brace and its use as an accepted treatment for knee OA is to be advocated for general use.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all criteria listed below will be considered to eligible for participation in the study:

* Patient, men and women, age 30 to 70 with knee OA not scheduled for surgery who understand the given information and are willing to participate in this study.
* Signed informed patient consent
* BMI < 35
* Knee pain for more than 3 month
* Patients with Knee OA Ahlbäck grade 1 and 2 and/or Kellgren-Lawrence 1 and 2
* Patient with arthroscopic OA but do not have regular grade 1 OA

Exclusion Criteria:

Patient presenting with any of the following will not be included in the study:

* prior major surgery to the same knee
* patients with a history of stroke or neurological or psychiatric decease that potentially could affect the perception of pain
* obesity (BMI > 35)
* active or suspected infection
* patients taking opioids or steroids
* patients suffering from rheumatoid arthritis or have a immunological depression
* patients with other severe medical problems that could affect the perioperative course
* the patient had an intraarticular steroid injection in the actual knee during the last 3 months
* Patient participating in a clinical trial

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | one year
  Standardized questionaire for knee problems, divided into 5 subscores of pain, symptoms, activity of daily living, sports/recreation and quality of life. Each subscore is presented from 0 (worst) to 100 (best).
Knee Society Score (KSS) | one year
  Standardized outcome measure for knee problems presented in two subgroups of KSS Score and KSS Function, presented on a range from 0 (worst) to 100 (best)
Visual Analogue Scale (VAS) | one year
  VAS is presented as a range from 0 (no pain) to 100 (worst possible pain)
EQ-5D | one year
  EQ-5D comprises two distinct self-report elements, providing three principal approaches to analysis(1) the EQ-5D profile: the patients' self reported health on the dimensions/levels of the descriptive system (2) the EQ-VAS: the patients' own global rating of their overall health, on a scale from 0 (worst possible health) to100 (best possible health)• Both types of data can be the focus of analysis, plus(3) Profiles can be summarized using 'value sets' (EQ-5DIndex) which reflect the preferences of the general public.

CONTACTS AND LOCATIONS:
Overall Officials: Soren Toksvig-Larsen, Ass prof, Principal Investigator — Orthopeadic Clinic Hassleholm
Locations (1):
- Orthopeadic Clinic Hässlehlm Hospital, Hässleholm, Skåne County, Sweden

REFERENCES:
- [Derived] Hjartarson HF, Toksvig-Larsen S. The clinical effect of an unloader brace on patients with osteoarthritis of the knee, a randomized placebo controlled trial with one year follow up. BMC Musculoskelet Disord. 2018 Sep 22;19(1):341. doi: 10.1186/s12891-018-2256-7. PMID 30243296